CLINICAL TRIAL: NCT06783400
Title: What Works to Prevent Violence Against Women and Girls: Impact at Scale: A Cluster Randomized Controlled Trial to Assess the Effectiveness of a Community-mobilisation Intervention to Prevent Violence Against Women in Malawi - SASA! Together
Brief Title: What Works - Malawi SASA! Together
Acronym: WW-M-SASA!
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Global Women's Institute (Unknown); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCR245830SASA
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Intimate Partner Violence (IPV); Norms, Social; Gender Inequitable Behavior
Keywords: intimate partner violence; gender; social norms; community mobilization; behavior change
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In control communities SASA! Together will not be implemented.
- SASA! Together (Experimental): The SASA! Together programme will be implemented in communities in this arm.
  Interventions: Behavioral: SASA! Together

INTERVENTIONS:
Behavioral: SASA! Together — SASA! Together is a community mobilisation approach that engages communities to create positive and sustainable changes around norms and behaviors that perpetuate violence against women. Some new features in this revision of SASA! include a distinct focus on IPV, including sexual decision-making; three strategies aligned to the socio-ecological model that reach across the whole community (individuals, groups, and institutions); and more support to get organisations and communities started and to sustain change.
  The evidence- and theory-based SASA! approach is grounded in: (1) benefits-based activism, (2) a gender-power analysis, (3) four phases of change (start, awareness, support, action) according to the stages of behaviour change, (4) holistic community engagement, (5) local activism, (6) community leadership, and (7) institutional strengthening.
  Arms: SASA! Together

SUMMARY:
Violence against women is complex and must be addressed at multiple levels, with leadership from women themselves on how to bring about positive change to free women and girls from daily experiences of violence and to promote their rights. It is in this context that the Pamodzi Kuthetsa Nkhanza (PKN) consortium will implement a programme to facilitate the prevention of intimate partner violence (IPV) in Malawi as one of the most common forms of VAW experienced in Malawi. The programme takes a whole community approach and uses gender transformative approaches at different levels of society to address the root causes of IPV. It will draw primarily on two existing, evidence-based prevention models, namely SASA! Together (community mobilisation model) and Moyo Olemekeza (MO) (gender norms and behaviour change and economic empowerment approach).

A cluster randomised controlled trial (cRCT) will evaluate the effectiveness of the PKN programme, assessing the effectiveness of the SASA! Together programme at shifting individual behaviours and reducing violence in intimate relationships while also tackling community norms that drive these forms of violence against women. The cRCT will also assess the added value of combining SASA! Together and a women's social and economic empowerment programme (MO) for most at-risk households.

This protocol focuses on the evaluation of the SASA! Together programme.

DETAILED DESCRIPTION:
According to the 2016 Malawi Demographic and Health Survey, 42% of ever-married women aged 15 - 49 have experienced spousal physical, sexual, or emotional violence by their current or most recent spouse, and a third (33%) of ever-married women experienced at least one of these forms of violence in the 12 months before the survey [1]. Overall, 41% of all women (whether they have ever been married or not) have experienced physical or sexual violence [1]. Despite these high levels of violence against women and girls (VAWG), there are a limited number of evidence-based interventions focused on preventing VAW in Malawi.

Violence against women must be addressed at multiple levels, with leadership from women themselves on how to bring about positive change to free women and girls from daily experiences of violence and to promote their rights. It is in this context that the Pamodzi Kuthetsa Nkhanza (PKN) consortium will implement a programme to facilitate the prevention of intimate partner violence (IPV) in Malawi. The programme takes a whole community approach and uses gender transformative approaches at different levels of society to address the root causes of IPV. It will draw primarily on two existing, evidence-based prevention models, namely SASA! Together and Moyo Olemekeza (MO).

This cRCT forms part of a broader mixed methods research design. Guided by the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework, the overall research design consists of five distinct components, all contributing to evidence on the efficacy of the programme and the contextual factors around the programme and its implementation that will guide the interpretation of the cRCT.

This protocol refers to the cRCT evaluation of SASA! Together only. Specifically, the cRCT aims to evaluate the community level impact of SASA! Together on experiences of IPV among women aged 18 - 49 in two districts in Malawi (Balaka and Lilongwe districts).

The specific aim for understanding the efficacy of the SASA! Together programme is:

1) To estimate the community-level causal impact of SASA! Together (compared to a control) on the primary and secondary outcomes among women and men aged 18 - 49 in Lilongwe and Balaka districts, Malawi.

The overall goal of this study is to add to the evidence base on effective, comprehensive interventions to reduce violence against women in Malawi.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18-49 who have ever been in an intimate (romantic) relationship.
* Living in selected Group Village Heads (GVHs) in Lilongwe or Balaka districts for at least a year. The specific Traditional Authorities (TAs) in Lilongwe are: Kalolo, Chimutu, Kabudula; The TAs in Balaka are: Msamala and Nyanyala.

Exclusion Criteria:

* Women and men younger than 18 years or older than 49 years old
* Women who have never had an intimate relationship.
* Not living in selected TAs and GVHs in Lilongwe or Balaka districts, or living in selected GVHs for less than one year
* Paid employees of the PKN programme (any element), including SASA! Together community activists who deliver the programme activities.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4800 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Indicator for Past year experience of any violence (physical, sexual, or emotional) from a partner (among women who have had an intimate partner in the past year) | 12 months
  Defining past year experience of intimate partner violence using the World Health Organization's "Multi-country study measure for intimate partner violence" module.
Acceptability of violence (personal belief; among men and women separately) | From time of implementation to endline assessment is 3 years
  Sum of indicators that the respondent agrees that a man/husband has a good reason to hit or beat his wife/partner if she (1) goes out without telling him; (2) she neglects the children; (3) she argues with him; (4) she refuses to have sex with him; (5) she burns the food; (6) he suspects that she has been unfaithful

SECONDARY OUTCOMES:
Indicator for Past year experience of physical violence from a partner (among women who have had an intimate partner in the past year) | 12 months
  An indicator equal to one if the respondent reports a partner perpetrated any of the following behaviors in the past 12 months: (i) Slapped you or thrown something at you (ii)Pushed or shoved you (iii) Hit you with his fist or with something else (iv) Kicked, dragged or beaten you (v) Choked or burnt you and (vi) Threatened you with, or actually used, a knife or other weapon against you
Indicator for Past year experience of sexual violence from a partner (among women who have had an intimate partner in the past year) | 12 months
  An indicator equal to one if the respondent reports a partner perpetrated any of the following behaviors in the past 12 months: (i) Physically forced you to have sexual intercourse (ii) Physically forced you to perform any other sexual acts (iii) Force you with threats to perform sexual acts
Indicator for Past year experience of emotional violence from a partner (among women who have had an intimate partner in the past year) | 12 months
  An indicator equal to one if the respondent reports a partner perpetrated any of the following behaviors in the past 12 months: (i) Insulted you or made you feel bad about yourself (ii) Destroyed things that are important to you (iii) Did things that made you feel scared or intimidated (iv) Threatened to harm you or someone you care about (v) Thrown you out of the house (vi) Taken away your phone or controlled how you use it
Indicator for Past year experience of economic violence from a partner (among women who have had an intimate partner in the past year) | 12 months
  An indicator equal to one if the respondent reports a partner perpetrated any of the following behaviors in the past 12 months: (i) Prohibits you from earning money (ii) Takes earnings from you against your will (iii) Refuses to give money for household expenses (iv) Keeps you from getting a loan (v) Not let you participate in deciding how the family finances are spend
Indicator for Past year experience of controlling behaviour from a partner (among women who have had an intimate partner in the past year) | 12 months
  An indicator equal to one if the respondent reports a partner perpetrated any of the following behaviors in the past 12 months: (i) Tries to stop you from meeting your friends (ii) Tries to limit contact with your family of birth (iii) Insists on knowing where you are at all times (iv) Gets jealous or angry if you talk with another man (v) Frequently accuses you of being unfaithful (vi) Checks your cellphone/WhatsApp logs/messages to see who you have called or messaged/who has called or messaged you
Index for Acceptability of intimate partner violence (among all women and men separately) | From time of implementation to endline assessment is 3 years
  This measure is a summation of the responses to each of 4 relationship attitudes, with a possible maximum score of 4. Higher scores will indicate more restrictive attitudes towards violence. Components are:
  * Indicator for Agrees that violence between husband and wife is a private matter and others should not intervene
  * Indicator for Agrees that a woman should tolerate violence to keep her family together
  * Indicator for Agrees that if a woman is raped, she has usually done something careless
  * Indicator for Agrees that if a woman doesn't physically fight back, you can't really call it rape
Index of Appropriate community response to women experiencing IPV in past year (among all women and men separately) | From time of implementation to endline assessment is 3 years
  This measure is a summation of two indicators:
  * Indicator witnessed/heard and helped when violence was happening between husbands and wives in the community
  * Indicator for was told and helped a woman in community told who experienced violence from her partner

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Legal Resources Center (WOLREC), Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual-level data sets
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Information will be made available upon request after primary manuscripts have been published